CLINICAL TRIAL: NCT05156398
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rimegepant in Migraine Prevention in Children and Adolescents ≥ 6 to <18 Years of Age
Brief Title: Efficacy and Safety Study of Rimegepant for the Preventative Treatment of Migraine in Pediatric Subjects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BHV3000-315; C4951009 (Other: Alias Study Number); 2021-005246-15 (EudraCT Number: CTIS (EU)); 2021-005246-15 (Registry Identifier: CTIS (EU)); 2024-512382-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-11-19; First posted 2021-12-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Migraine; Migraine prevention; Phonophobia; Photophobia; Nausea; Pediatric migraine; Adolescent migraine
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rimegepant / BHV3000 (Active Comparator): Rimegepant 75mg or 50mg (2 X 25mg) ODT
  Interventions: Drug: Rimegepant
- Matching Placebo (Placebo Comparator): Matching placebo 75mg or 50mg (2 X 25mg) ODT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75mg or 50mg (2 X 25mg) ODT
  Other Names: BHV3000
  Arms: Rimegepant / BHV3000
Drug: Placebo — Matching placebo 75mg or 50mg (2 X 25mg) ODT
  Other Names: Matching Placebo
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of rimegepant to placebo as a preventative treatment for migraine in children and adolescents ≥ 6 to <18 years with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least a 6 month history of migraine (with or without aura) and including the following:

   1. 14 or less headache days per month during the 3 month period prior to the Screening Visit
   2. 6 or more migraine days during the Observation Period
   3. 14 or less headache days during the Observation Period
   4. Pediatric Migraine Disability Assessment Scale (PedMIDAS) Disability Score of >10 to ≤50, indicating mild (score of 11 to 30) or moderate (score of 31 to 50) disruption in daily activities, as assessed at the Baseline (Randomization) Visit
   5. Ability to verbally distinguish migraine attacks from tension/cluster or other types of headaches
   6. Migraine attacks, on average, lasting 4 - 72 hours if untreated
   7. Subjects on prophylactic migraine medication are permitted to remain on therapy if the dose has been stable for at least 3 months (12 weeks) prior to the Screening Phase, and the dose is not expected to change during the course of the study. 2) Male and female subjects ≥ 6 to <18 years; subjects must be less than 18 at the time of signing assent / consent.

      3)Subjects must have a weight of ≥40 kg (child cohort requirement ≥15 kg) at the Screening Visit.

Exclusion Criteria:

1. Subjects with a history of basilar migraine, cluster headaches, or hemiplegic migraine
2. The subject has a continuous migraine (defined as an unrelenting headache) within 1 month prior to Screening Visit.
3. The subject has a history or diagnosis of complications of migraine
4. The subject has a confounding and clinically significant pain syndrome that may interfere with the subject's ability to participate in this study.
5. The subject has any current psychiatric condition that is uncontrolled and/or untreated for a minimum of 6 months prior to the Screening Visit. Subjects with a lifetime history of psychosis and/or mania are excluded.
6. History of suicidal behavior or the subject is at risk of self-harm or harm to others.
7. History of major psychiatric disorder.
8. The subject has a current diagnosis or history of substance abuse
9. The subject has a history of moderate or severe head trauma or other neurological disorder (including seizure disorder) or systemic medical disease that is, in the investigator's opinion, likely to affect central nervous system functioning.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 640 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2031-11-29 (Estimated); Study Completion 2032-11-27 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean number of migraine days per month as measured over the 12-week double-blind phase of the study in adolescents with episodic migraine | 3 months (12 weeks)
  Reduction from baseline in mean number of migraine days per month

SECONDARY OUTCOMES:
Achievement of at least a 50% reduction from baseline in mean monthly migraine days over the course of the double-blind phase in adolescents with episodic migraine | 3 months (12 weeks)
Change from baseline in the mean number of migraine days per month in the first 4 weeks (Weeks 1 through 4) of the double-blind treatment phase in adolescents with episodic migraine. | Weeks 1 through 4 of treatment
The mean change from baseline in the Pediatric Quality of Life (PedsQL™) total score at Week 12 of the double-blind treatment phase in adolescents with episodic migraine. | Total score at week 12
Change from baseline in the mean number of migraine days per month over the entire course of the double-blind treatment phase in children and children and adolescents combined with episodic migraine. | 3 months (12 weeks)
Change from baseline on the proportion of subjects that have at least a 50% reduction in the mean number of moderate to severe migraine days per month. | 3 months (12 weeks)
  Measured over the entire course of the double-blind treatment phase in children and children and adolescents combined with episodic migraine.
Compare the use of acute migraine-specific medications (triptans) based on the change from baseline in monthly acute migraine specific medication days. | 3 months (12 weeks)
  Measured in each month and over the course of the entire double-blind treatment phase in adolescents, children and adolescents and children combined.
Evaluate the safety and tolerability of rimegepant as a preventative treatment for migraine in children and adolescents. | 72 Weeks
  This will be evaluated by the number of subjects with treatment related adverse events by severity.
Evaluate the frequency of hepatic-related adverse events in subjects treated with rimegepant. | 72 Weeks
  Measured by discontinuations in treated subjects due to elevated liver function tests.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (91):
- United States (52):
  - The Belinga Clinic, Fort Smith, Arkansas
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Velocity Clinical Research San Diego, La Mesa, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Meridian Clinical Research, LLC, Washington D.C., District of Columbia
  - Accel Research Sites Network - Edgewater Clinical Research Unit, Edgewater, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - New Med Research, Inc, Hollywood, Florida
  - Complete Health Research, Ormond Beach, Florida
  - D&H Tamarac Research Center LLC, Tamarac, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Extraordinary Family Healthcare, Snellville, Georgia
  - Renew Health Clinical Research LLC, Snellville, Georgia
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Diamond Headache Clinic, Chicago, Illinois
  - Nola Research Works, LLC, New Orleans, Louisiana
  - Safe Haven Clinical Research, Clinton, Mississippi
  - Roy Blunt NextGen Precision Health Building, Columbia, Missouri
  - University of Missouri Health Care - Investigation Pharmacy, Columbia, Missouri
  - University of Missouri-Clinical and Translational Sciences Unit, Columbia, Missouri
  - Velocity Clinical Research, Inc., Grand Island, Nebraska
  - Papillion Research Center/CCT Research, Papillion, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Institute for Clinical Research, LLC, Fayetteville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Coastal Pediatric Research, Charleston, South Carolina
  - Tribe Clinical Research LLC, Greenville, South Carolina
  - Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota
  - Avera Research Institute, Sioux Falls, South Dakota
  - Avera Medical Group Pediatrics - Dawley Farm, Sioux Falls, South Dakota
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Alina Clinical Trials, LLC., Dallas, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - DM Clinical Research - Cy Fair, Houston, Texas
  - SCLA Management - Drop Box, Houston, Texas
  - SCLA Management Office, Houston, Texas
  - NeuroCare Plus, Houston, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - DCT-McAllen Primary Care Research, LLC dba Discovery Clinical Trials, McAllen, Texas
  - DCT-Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - DM Clinical Research (Administrative Office Only), Tomball, Texas
  - Victoria Clinical Research Group, Victoria, Texas
  - Meridian Clinical Research, LLC, Portsmouth, Virginia
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada
- France (3):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Hopital des Enfants, Toulouse
- Italy (7):
  - UOSVD Centro Epilessia ed EEG dellEta Evolutiva, Bari, BARI / Puglia
  - Spedali Civili di Brescia, Brescia, Brescia/lombardy
  - Sapienza Universita di Roma Polo Pontino - ICOT, Headache clinic, Latina, Latina/lazio
  - Ospedale Pediatrico Bambino Gesu, Rome, Lazio
  - IRCCS San Raffaele, Rome, Lazio
  - Istituto Neurologico "Carlo Besta" Fondazione IRCCS, Milan, Lombardy
  - U.O. Neuropsichiatria Infantile, IRCCS Fondazione Mondino, Pavia, Lombardy
- Japan (14):
  - Jinnouchi Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - Hikita Pediatric Clinic, Kiryu-shi, Gunma
  - Konan Medical Center, Higashinada-ku Kobe-shi, Hyōgo
  - Yamaguchi Clinic, Nishinomiya-shi, Hyōgo
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Tanaka Neurosurgery & Headache Clinic, Kagoshima, Kagoshima-ken
  - Atago Hospital, Kochi, Kochi
  - Sendai Headache and Neurology Clinic, Taihaku-ku Sendai-shi, Miyagi
  - Tennouji Dai Brain Clinic, Abeno-ku Osaka-shi, Osaka
  - Tominaga Clinic, Naniwa-ku, Osaka
  - Saitama Neuropsychiatric Institute, Chuo-ku Saitama-shi, Saitama
  - Tokyo Headache Clinic, Shibuya-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - LIAC Hiroshima City Hospital Organization Hiroshima City Hiroshima Citizens Hospital, Hiroshima
- Poland (8):
  - Clinical Research Center Sp. z o.o. MEDIC-R Sp. k., Poznan, Greater Poland Voivodeship
  - Wojewodzki Specjalistyczny Szpital Dzieciecy, Krakow, Lesser Poland Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin, Lublin Voivodeship
  - MTZ Clinical Research Powered by Pratia, Warsaw, Masovian Voivodeship
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice, Silesian Voivodeship
  - Neurologia Slaska Centrum Medyczne, Katowice, Silesian Voivodeship
  - Next Stage Sp. Z o.o., Warsaw, WOJ. Mazowieckie
- Spain (6):
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital Clinico Universitario de Valladolid (HCUV), Valladolid, Castille and León
  - Hospital Alvaro Cunqueiro, Vigo, Galicia
  - Instituto de Investigaciones del Sueno, Madrid
  - Virgen del Rocio Hospital, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-315